CLINICAL TRIAL: NCT04201418
Title: A Phase 4 Multicenter Observational Study to Evaluate the Effectiveness of Patisiran in Patients With Polyneuropathy of Hereditary Transthyretin-Mediated (ATTRv) Amyloidosis With a V122I or T60A Mutation
Brief Title: A Multicenter Observational Study to Evaluate the Effectiveness of Patisiran in Patients With Polyneuropathy of ATTRv Amyloidosis With a V122I or T60A Mutation
Status: Completed | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTR02-012
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Hereditary Transthyretin-mediated (ATTRv) Amyloidosis; Polyneuropathy
Keywords: Valine to isoleucine substitution at position 122; V122I; Threonine to alanine substitution at position 60; T60A; Familial Amyloid Polyneuropathies; ATTR; Transthyretin amyloidosis; Transthyretin; Amyloidosis; TTR-mediated Amyloidosis; RNAi therapeutic; FAP; Polyneuropathies; Amyloid neuropathies; Amyloid neuropathies, familial; Amyloidosis, familial; Peripheral nervous system diseases; Nervous system diseases; TTR; Neuromuscular diseases; Proteostasis deficiencies; Metabolic diseases; Heredodegenerative disorders, nervous system; Neurodegenerative diseases; Genetic diseases, inborn; Metabolism, inborn errors; ATTRv
MeSH Terms: conditions — Amyloidosis; Polyneuropathies; Amyloid Neuropathies, Familial; Amyloidosis, Hereditary, Transthyretin-Related; Amyloid Neuropathies; Amyloidosis, Familial; Peripheral Nervous System Diseases; Nervous System Diseases; Neuromuscular Diseases; Proteostasis Deficiencies; Metabolic Diseases; Heredodegenerative Disorders, Nervous System; Neurodegenerative Diseases; Genetic Diseases, Inborn; Metabolism, Inborn Errors | interventions — patisiran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Patisiran Prospective Cohort: Patients who are naive to patisiran at study enrollment with the intention to initiate commercial patisiran therapy.
  Interventions: Drug: Patisiran
- Patisiran Mixed Cohort: Patients who are currently on commercial patisiran therapy for less than 12 months at study enrollment.
  Interventions: Drug: Patisiran
- Patisiran Retrospective Cohort: Patients who have been on commercial patisiran therapy for at least 12 months prior to study enrollment, regardless of current treatment status at enrollment.
  Interventions: Drug: Patisiran

INTERVENTIONS:
Drug: Patisiran — Patisiran-lipid complex injection, for intravenous use
  Other Names: ONPATTRO; ALN-TTR02

SUMMARY:
To evaluate the effectiveness of patisiran in patients with ATTRv amyloidosis with polyneuropathy who have a V122I or T60A mutation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ATTRv amyloidosis with polyneuropathy, with a documented V122I or T60A mutation
* PND score of I-IIIB at baseline.
* Exposure to commercial patisiran in one of the 3 cohorts:

  * Prospective Cohort: Naive to patisiran treatment at the time of enrollment with intention to initiate treatment with patisiran.
  * Mixed cohort: Currently on commercial patisiran therapy for less than 12 months at study enrollment.
  * Retrospective cohort: Exposed to commercial patisiran treatment for at least 12 months prior to study enrollment, regardless of current treatment status at enrollment.

Exclusion Criteria:

* New York Heart Association (NYHA) heart failure classification ≥3
* Karnofsky Performance Status (KPS) <60%
* Unstable congestive heart failure (CHF)
* Known primary amyloidosis (AL) or leptomeningeal amyloidosis
* Prior major organ transplant
* Previously received patisiran
* Previous treatment with a TTR silencing therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ATTRv amyloidosis with polyneuropathy who have a V122I or T60A mutation
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Stable or Improved Polyneuropathy Disability (PND) Score at 12 Months Relative to Baseline | Baseline, Month 12
  PND Scores: Stage 0=No symptoms, Stage 1=Sensory disturbances but preserved walking capability, Stage 2=Impaired walking capacity, but ability to walk without a stick or crutches, Stage 3A/B=Walking with the help of 1 or 2 sticks or crutches, Stage 4=confined to wheel chair or bedridden.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (25):
- United States (25):
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, San Diego, California
  - Clinical Trial Site, Aurora, Colorado
  - Clinical Trial Site, Farmington, Connecticut
  - Clinical Trial Site, Jacksonville, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Braselton, Georgia
  - Clinical Trial Site, Macon, Georgia
  - Clinical Trial Site, Chicago, Illinois
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Detroit, Michigan
  - Clinical Trial Site, Jackson, Mississippi
  - Clinical Trial Site, Kansas City, Missouri
  - Clinical Trial Site, Omaha, Nebraska
  - Clinical Trial Site, Chapel Hill, North Carolina
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Allentown, Pennsylvania
  - Clinical Trial Site, Bethlehem, Pennsylvania
  - Clinical Trial Site, Lancaster, Pennsylvania
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Germantown, Tennessee
  - Clinical Trial Site, Austin, Texas
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No